CLINICAL TRIAL: NCT03760770
Title: Riboflavin at 4ºC for the Management of Pain After Crosslinking for Keratoconus Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEI-2018/10/01
Record Dates: First submitted 2018-11-28; First posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Keratoconus; Crosslinking
Keywords: Crosslinking; Keratoconus; Cold; Pain
MeSH Terms: conditions — Keratoconus; Common Cold; Pain | interventions — Corneal Cross-Linking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Riboflavin at 4ºC (Experimental): patients treated with Riboflavin at 4ºC in crosslinking (cases).
  Interventions: Procedure: corneal collagen crosslinking
- Riboflavin at room temperature (Experimental): patients treated with Riboflavin at room temperature in crosslinking (controls)
  Interventions: Procedure: corneal collagen crosslinking

INTERVENTIONS:
Procedure: corneal collagen crosslinking — Crosslinking in patients with progressive keratoconus.
  Other Names: No Cold riboflavin (Riboflavin at room temperature); Cold riboflavin (Riboflavin at 4ºC)

SUMMARY:
Background: The objective of corneal collagen crosslinking (CXL) is to increase the binding of intrafibrillary and interfibrillary covalent bonds to improve the mechanical stability of the cornea and thus to stop the progression of corneal ectasias. Although the vast majority of studies have described pain after photorefractive keratectomy (PRK), the pathophysiological principle of pain is similar in CXL. From the anatomical point of view, the corneal epithelium is the most densely innervated and sensitive surface of the body, being 300-600 times greater than in the skin. The pain after CXL comes from several routes, the process begins with the epithelial rupture that generates exposure of the nerve endings, induces apoptosis and necrosis of the epithelial cells. Subsequently an inflammatory cascade is initiated in which the different cytokines stimulate the nerve terminals. Inflammatory mediators also activate the ion channels in the nerve membrane, and this process continues until the epithelium heals. Additionally, exposure to UVA rays can also cause nerve damage. The effect of local cold for pain management has already been reported in PRK. By cooling the cornea, the release of chemical mediators and inflammation can be reduced. In the CXL radiation is transformed into several forms of energy: fluorescent radiation, chemical energy and, to a small extent, heat. The CXL process is energetically comparable to photosynthesis, in which the radiation energy is transformed into chemical energy (glucose) with the help of pigments (chlorophyll). The thermal effect is negligible in the photochemical method of CXL. Justification: No method for the control of pain after crosslinking is considered ideal or universally accepted, the importance of this study lies in looking for an additional tool to reduce the most common postoperative complaint in a highly performed procedure worldwide. Hypothesis: The application of riboflavin at 4oC reduces the pain assessment after the CXL. Purpose: to evaluate the effect of the application of riboflavin at 4oC in the assessment of postoperative pain in patients undergoing CXL. Materials and methods: Prospective and interventional clinical study in patients older than 18 years with a diagnosis of keratoconus who underwent CXL, in the cornea and refractive surgery service of the Ophthalmology institute Fundación Conde de Valenciana.

ELIGIBILITY:
Inclusion Criteria:

* patients of any gender
* older than 18 years
* diagnosis of keratoconus who require management with crosslinking in both eyes for evidence of progression.

Exclusion Criteria:

* crosslinking without removal of epithelium or unilateral crosslinking.
* patients with other ocular conditions different from keratoconus.
* cognitive disability that limits the compression of the pain test as Down syndrome, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Change pain perception in patients undergoing crosslinking with riboflavin at 4ºC | 2 postoperative hours and from day 1 to 5 postoperative.
  A previously validated numerical pain scale questionnaire was applied. Patients are asked to indicate their pain intensity on a scale of 0 to 10, explaining that 0 does not represent pain at all and 10 is a severe and disabling pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de oftalmología conde de Valenciana, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Spadea L, Salvatore S, Paroli MP, Vingolo EM. Recovery of corneal sensitivity after collagen crosslinking with and without epithelial debridement in eyes with keratoconus. J Cataract Refract Surg. 2015 Mar;41(3):527-32. doi: 10.1016/j.jcrs.2014.06.030. Epub 2015 Jan 30. PMID 25648281
- [Result] Mencucci R, Mazzotta C, Rossi F, Ponchietti C, Pini R, Baiocchi S, Caporossi A, Menchini U. Riboflavin and ultraviolet A collagen crosslinking: in vivo thermographic analysis of the corneal surface. J Cataract Refract Surg. 2007 Jun;33(6):1005-8. doi: 10.1016/j.jcrs.2007.03.021. PMID 17531694
- [Result] Garcia R, de Andrade DC, Teixeira MJ, Nozaki SS, Bechara SJ. Mechanisms of Corneal Pain and Implications for Postoperative Pain After Laser Correction of Refractive Errors. Clin J Pain. 2016 May;32(5):450-8. doi: 10.1097/ajp.0000000000000271. PMID 27504514
- [Result] Woreta FA, Gupta A, Hochstetler B, Bower KS. Management of post-photorefractive keratectomy pain. Surv Ophthalmol. 2013 Nov-Dec;58(6):529-35. doi: 10.1016/j.survophthal.2012.11.004. PMID 24160728
- [Result] Xia Y, Chai X, Zhou C, Ren Q. Corneal nerve morphology and sensitivity changes after ultraviolet A/riboflavin treatment. Exp Eye Res. 2011 Oct;93(4):541-7. doi: 10.1016/j.exer.2011.06.021. Epub 2011 Jul 13. PMID 21763309
- [Result] Kitazawa Y, Maekawa E, Sasaki S, Tokoro T, Mochizuki M, Ito S. Cooling effect on excimer laser photorefractive keratectomy. J Cataract Refract Surg. 1999 Oct;25(10):1349-55. doi: 10.1016/s0886-3350(99)00207-2. PMID 10511934
- [Result] Raiskup F, Spoerl E. Corneal crosslinking with riboflavin and ultraviolet A. I. Principles. Ocul Surf. 2013 Apr;11(2):65-74. doi: 10.1016/j.jtos.2013.01.002. Epub 2013 Jan 24. PMID 23583042
- [Result] Sharif R, Bak-Nielsen S, Hjortdal J, Karamichos D. Pathogenesis of Keratoconus: The intriguing therapeutic potential of Prolactin-inducible protein. Prog Retin Eye Res. 2018 Nov;67:150-167. doi: 10.1016/j.preteyeres.2018.05.002. Epub 2018 Jul 13. PMID 29758268
- [Result] Galvis V, Tello A, Carreno NI, Berrospi RD, Nino CA. Risk Factors for Keratoconus: Atopy and Eye Rubbing. Cornea. 2017 Jan;36(1):e1. doi: 10.1097/ICO.0000000000001052. No abstract available. PMID 27755195
- [Result] Godefrooij DA, de Wit GA, Uiterwaal CS, Imhof SM, Wisse RP. Age-specific Incidence and Prevalence of Keratoconus: A Nationwide Registration Study. Am J Ophthalmol. 2017 Mar;175:169-172. doi: 10.1016/j.ajo.2016.12.015. Epub 2016 Dec 28. PMID 28039037
- [Result] Ghanem VC, Ghanem RC, de Oliveira R. Postoperative pain after corneal collagen cross-linking. Cornea. 2013 Jan;32(1):20-4. doi: 10.1097/ICO.0b013e31824d6fe3. PMID 22547128
- [Result] Wollensak G, Spoerl E, Seiler T. Riboflavin/ultraviolet-a-induced collagen crosslinking for the treatment of keratoconus. Am J Ophthalmol. 2003 May;135(5):620-7. doi: 10.1016/s0002-9394(02)02220-1. PMID 12719068
- [Result] Peyman A, Nouralishahi A, Hafezi F, Kling S, Peyman M. Stromal Demarcation Line in Pulsed Versus Continuous Light Accelerated Corneal Cross-linking for Keratoconus. J Refract Surg. 2016 Mar;32(3):206-8. doi: 10.3928/1081597X-20160204-03. PMID 27027629
- [Result] Kymes SM, Walline JJ, Zadnik K, Sterling J, Gordon MO; Collaborative Longitudinal Evaluation of Keratoconus Study Group. Changes in the quality-of-life of people with keratoconus. Am J Ophthalmol. 2008 Apr;145(4):611-617. doi: 10.1016/j.ajo.2007.11.017. Epub 2008 Jan 28. PMID 18226798
- [Result] Lichtinger A, Purcell TL, Schanzlin DJ, Chayet AS. Gabapentin for postoperative pain after photorefractive keratectomy: a prospective, randomized, double-blind, placebo-controlled trial. J Refract Surg. 2011 Aug;27(8):613-7. doi: 10.3928/1081597X-20110210-01. Epub 2011 Feb 28. PMID 21366172
- [Result] Spadea L, Tonti E, Vingolo EM. Corneal stromal demarcation line after collagen cross-linking in corneal ectatic diseases: a review of the literature. Clin Ophthalmol. 2016 Sep 19;10:1803-1810. doi: 10.2147/OPTH.S117372. eCollection 2016. PMID 27695286
- [Result] Yam JC, Chan CW, Cheng AC. Corneal collagen cross-linking demarcation line depth assessed by Visante OCT After CXL for keratoconus and corneal ectasia. J Refract Surg. 2012 Jul;28(7):475-81. doi: 10.3928/1081597X-20120615-03. PMID 22767165